CLINICAL TRIAL: NCT01712152
Title: Myocardial Involvement in Carriers of Duchenne Muscular Dystrophy: An MRI-study
Status: Completed | Type: Observational
Sponsor: Hospital Rudolfstiftung (Other)
Collaborators: Oesterreichische Muskelforschung (Unknown)
Responsible Party: Principal Investigator, Paul Wexberg,MD, Priv.-Doz., Hospital Rudolfstiftung
Other Study IDs: EK 11-228- 0112
Record Dates: First submitted 2012-10-19; First posted 2012-10-23 (Estimated); Last update posted 2016-10-04 (Estimated); Status verified 2016-10

CONDITIONS: Carrier of Duchenne Muscular Dystrophy
Keywords: Duchenne muscular dystrophy; carrier; cardiac MRI; myocardial fibrosis; female
MeSH Terms: conditions — Muscular Dystrophy, Duchenne

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Carriers of Duchenne muscular dystrophy (DMD) often have no severe symptoms of the scelet muscles, but they may develop a poor heart function due to the involvement of the heart muscle. Ultrasound of the heart is recommended, but it can detect a cardiac affection only after the heart has already become weaker. Cardiac magnetic resonance tomography can detect myocardial fibrosis already at preserved heart function and may facilitate early therapy. In our study, diagnosed carriers of DMD will undergo examinations of the heart by blood tests, EKG, heart ultrasound and magnetic resonance at enrollment and after one year in order to assess the extent of cardiac affection and its association with the clinical development.

ELIGIBILITY:
Inclusion Criteria:

genetic and/or histological identification as a carrier of DMD age above 18 years able and willing to conform to the requirements of the study provided written informed consent exclusion of pregnancy in women of childbearing potential

Exclusion Criteria:

Claustrophobia Excessive obesity to an extent where CMR cannot be performed Chronic renal failure with a GFR <30 ml/min/1,73m² Implanted pacemakers/defibrillators Severe arrhythmia Inability to cooperate during the CMR Known intolerance to gadolinium Positive pregnancy test Unable or unwilling to conform to the study protocol

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: data base of carriers of Duchenne muscular dystrophy
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2012-10; Primary Completion 2014-04 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
T1 mapping | 1 year
  T1 mapping by MOLLI sequences will be performed and compared between study entry and one year follow-up

SECONDARY OUTCOMES:
left ventricular function | 1 year
  left ventricular function on MRI will be compared between study entry and one year follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Paul Wexberg, MD, Study Director — Hospital Rudolfstiftung
Locations (1):
- 2nd Medical Dept., Rudolfstiftung, Vienna, Austria

REFERENCES:
- [Derived] Wexberg P, Avanzini M, Mascherbauer J, Pfaffenberger S, Freudenthaler B, Bittner R, Bernert G, Weidinger F. Myocardial late gadolinium enhancement is associated with clinical presentation in Duchenne muscular dystrophy carriers. J Cardiovasc Magn Reson. 2016 Sep 22;18(1):61. doi: 10.1186/s12968-016-0281-y. PMID 27660108